CLINICAL TRIAL: NCT02947620
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of Metformin/Atorvastatin Combination Therapy in Subjects With Type II Diabetes and Dyslipidemia
Brief Title: Metformin/Atorvastatin Combination Therapy in Subjects With Type II Diabetes and Dyslipidemia (Phase 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_MA001
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2016-10

CONDITIONS: Type II Diabetes; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Metformin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Metformin/Atorvastatin (Active Comparator): Metformin/Atorvastatin, QD
  Interventions: Drug: Metformin/Atorvastatin 1500mg/40mg, QD
- Metformin (Placebo Comparator): Metformin, QD
  Interventions: Drug: Atorvastatin 40mg, QD
- Atorvastatin (Placebo Comparator): Atorvastatin, QD
  Interventions: Drug: Metformin 1500mg, QD

INTERVENTIONS:
Drug: Metformin/Atorvastatin 1500mg/40mg, QD
  Arms: Metformin/Atorvastatin
Drug: Metformin 1500mg, QD
  Arms: Atorvastatin
Drug: Atorvastatin 40mg, QD
  Arms: Metformin

SUMMARY:
A Multi-center, Randomized, double-blind, active-controlled, phase 3 trial to evaluate the safety and efficacy of Metformin/Atorvastatin in subjects with Type II Diabetes and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Dyslipidemia and Type II Diabetes
* 19 years later, men and women under the age of 80

Exclusion Criteria:

* Pregnant women, nursing mothers or subject who does not agree to assigned contraception in the study
* Subject with type I Diabetes
* Subject with hypertension which does not controlled by treatment(have blood pressure > 180/110mmHg)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-08; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Change from baseline at 16 weeks
  Change in HbA1c after 16 weeks, relative to baseline, between the combination of Metformin 1500 mg and Atorvastatin 40 mg compared to Atorvastatin 40 mg alone
Change in LDL Cholesterol | Change from baseline at 16 weeks
  Change in low-density lipoprotein cholesterol (LDL-C) after 16 weeks, relative to baseline, between Metformin 1500 mg alone and the combination of Metformin 1500 mg and Atorvastatin 40 mg

SECONDARY OUTCOMES:
Change in LDL-C | Baseline and 16 weeks
  Change in LDL-C after 16 weeks, relative to baseline, between Atorvastatin 40 mg and the combination of Metformin 1500 mg and Atorvastatin 40 mg
Change in HbA1c | Baseline and 16 weeks
  Change in HbA1c after 16 weeks, relative to baseline, between Metformin 1500 mg alone and the combination of Metformin 1500 mg and Atorvastatin 40 mg
Percentage of subjects reaching the LDL-C treatment goal defined by the NCEP ATP III guideline (<100mg/dL) after 16 weeks of treatment with investigational products | 16 weeks
Percentage of subjects reaching HbA1c <7.0% and <6.5% after 16 weeks of treatment with investigational products | 16 weeks
Change in LDL-C and the associated rate of change after 4, 8, and 12 weeks of treatment with investigational products compared to baseline | Baseline, 4 weeks, 8 weeks and 12 weeks
Change in LDL-C after 16 weeks, relative to baseline, in subjects treated with investigational products | Baseline and 16 weeks
Change in lipid variables and the associated rate of change | Baseline, 4 weeks, 8 weeks and 12 weeks and 16 weeks
  Change in lipid variables (HDL-C, TG, TC, non-HDL cholesterol, Apolipoprotein A1, Apolipoprotein B) and the associated rate of change after 4, 8, 12, and 16 weeks of treatment with investigational products compared to baseline
Change in average fasting plasma glucose (FPG) after 4, 8, 12, and 16 weeks of treatment with investigational products compared to baseline | Baseline, 4 weeks, 8 weeks and 12 weeks and 16 weeks
Change in Insulin, HOMA-β, HOMA-IR after 4, 8, 12, and 16 weeks of treatment with investigational products compared to baseline. | Baseline, 4 weeks, 8 weeks and 12 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea